CLINICAL TRIAL: NCT02816476
Title: A Multicentre Open Label Phase II Study of Daratumumab in AL Amyloidosis Patients Not in VGPR or Better
Brief Title: Daratumumab Therapy for Patients With Refractory or Relapsed AL Amyloidosis
Acronym: AMYDARA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I15015/AMYDARA
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daratumumab (Experimental): Patient will receive Daratumumab every week for the first 2 cycles then every 2 weeks from cycle 3 through cycle 6.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab

SUMMARY:
This is a Phase II, single-arm, multicentre study of Daratumumab (16mg/kg IV route) in adult patients with Light-Chain (AL) Amyloidosis who are not in VGPR or better after previous treatment. A sample size of 40 patients who meet all eligibility criteria will be enrolled to receive study treatment. Patients will receive treatment until either disease progression or toxicity has occurred with a maximum planned of six 28-day cycles.

Daratumumab will be administrated every week for the first 2 cycles then. every 2 weeks from cycle 3 through cycle 6.

Patients will also receive best supportive care (BSC) to mitigate Daratumumab side-effects, and to address underlying Amyloidosis, including blood product transfusions, antimicrobials, and (as appropriate) growth factors including granulocyte colony-stimulating factors for neutropenia, erythropoietin for anaemia, and/or transfusions for thrombocytopenia

DETAILED DESCRIPTION:
Systemic AL amyloidosis is a rare disease caused by the deposition of misfolded monoclonal immunoglobulin free light chains (FLC) in various tissues and organs. It is usually associated with a clonal plasma cell dyscrasia with a low tumour burden. Treatment of AL amyloidosis relies mainly on chemotherapy aimed at suppressing the underlying plasma cell clone secreting monoclonal FLC. The organ responses and the survival are greatly influenced by the degree of hematological response evaluated by the decrease in serum FLC that has been the principal endpoint in recent trials in AL amyloidosis. The goal of treatment is to reach at least a very good partial response (VGPR) defined as a difference between the involved FLC and the normal <40 mg/l.

Over the last 2 years, Daratumumab, a novel, high-affinity, therapeutic, human monoclonal antibodies (mAb) that specifically recognizes the CD38 epitope has emerged as a breakthrough targeted therapy for patients with myeloma. Taking into account that, in 90% of AL patients, the monoclonal cells producing amyloidogenic FLC are Cluster of Differentiation 38 (CD38) expressing plasma cells Daratumumab should be a promising treatment in AL amyloidosis.

The study will consist of 4 steps:

* A 21 day screening period This period start with screening visit which may occurs up to 21 days before the first study drug administration. After signature of the informed consent form, procedures will be performed to ensure patient meet all inclusion/exclusion criteria and document health status to receive study treatment. These assessments will include quality of life questionnaires
* A treatment period Patient eligible to enter the study will receive 6 cycles of 28 days of intra venous Daratumumab. During cycles 1 and 2, Daratumumab will be administered weekly at days 1, 8, 15, and 22 then from cycles 3 to 6, Daratumumab will be administered every two weeks at days 1 and 15. Patient will have assessments at the ignition of a new cycle to document haematological and organs response and intra cycle to watch for toxicities.
* An end of study visit (when PD or unacceptable adverse events occurs, or planned end of study visit). Study procedures will be performed at 28 days (± 15) after the last dose of study medication for all patients, including early termination patients.
* Followup period After treatment discontinuation, followup will be made to the patient every 3 months for at least 1 year to inquire about the patient's hematological and organ status, general health, and information on any new medical events.

DOSING REGIMEN

Daratumumab. Six 28-day cycles, 16 mg/kg administered by IV route, During cycle 1 and 2, Daratumumab will be administered weekly at days 1, 8, 15, and 22

For cycles 3 to 6, Daratumumab will be administered every other week at days 1 and 15

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >18 years of age
2. Histologic diagnosis of AL amyloidosis
3. Genetic testing must be negative for transthyretin mutations
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
5. Patients should have received at least one line with an alkylating agent and/or a proteasome inhibitor and dexamethasone and not be in VGPR or CR at the time of inclusion
6. Measurable hematologic disease:
7. Symptomatic organ involvement
8. Wash-out period of at least 4 weeks from previous antitumor therapy or any investigational treatment or 5 half-lives from previous antibodies, whichever is longer,
9. Adequate bone marrow function prior to 1st drug intake
10. Adequate organ function defined as:
11. Women with childbearing potential must be practicing one of the effective methods of birth control
12. A man who has not had a vasectomy and who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control
13. Only patients who are informed of the investigational nature of this study and sign and give written informed consent

Exclusion Criteria:

1. Amyloid-specific syndrome, such as carpal tunnel syndrome or skin purpura as the only evidence of disease. The finding of isolated vascular amyloid in a bone marrow biopsy specimen or in a plasmacytoma is not indicative of systemic amyloidosis
2. Isolated soft tissue involvement
3. Presence of non-AL amyloidosis
4. Bone marrow plasma cells >30% on bone marrow aspirate at screening
5. Cardiac mayo stage IIIb disease.
6. Repetitive ventricular arrhythmias on 24h Holter ECG despite anti-arrhythmic treatment, except if a pacemaker has been implanted.
7. Chronic atrial fibrillation
8. Supine systolic blood pressure <100 mmHg
9. Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of any component of the treatment regimen. Or, subject is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of any component of the treatment regimen
10. Clinically overt multiple myeloma with lytic bone lesions
11. Patients with uncontrolled infection or active malignancy
12. Any uncontrolled or severe cardiovascular or pulmonary disease
13. Subjects with psychiatric illnesses or social situations that would preclude them understanding the informed consent, study compliance or the ability to tolerate study procedures and/or study therapy
14. Subjects with known chronic obstructive pulmonary disease (COPD)
15. Subject has known moderate or severe persistent asthma within the past 2 years
16. Previous anti-CD38 therapy
17. Hypersensitivity to Dexamethasone that would prohibit treatment with study therapy
18. Known positive for HIV or active hepatitis B or C
19. Refusal to consent or protected by legal regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | After 6 cycles treatment (6 months).
  Overall Response Rate (CR+VGPR) at the completion of 6 cycles of Daratumumab using the new response criteria (J Clin Oncol, 2012. 30(36): p. 4541-9.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE V4.03. | Every month during 1 year

CONTACTS AND LOCATIONS:
Locations (10):
- France (9):
  - CHU d'Angers, Angers
  - CHU de Caen, Caen
  - CHU de Limoges, Limoges
  - CHU de Lyon Sud, Lyon
  - APHP - Necker, Paris
  - APHP - Saint Antoine, Paris
  - APHP - Saint Louis, Paris
  - CHU Poitiers, Poitiers
  - CHU de Rennes, Rennes
- Amyloidosis Research and Treatment Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No